CLINICAL TRIAL: NCT06705621
Title: Management and Clinical Outcome of Neonatal Arrhythmias in Assuit University Children's Hospital
Brief Title: Management and Clinical Outcome of Neonatal Arrhythmias
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manar Abdel-menem Fouad, 71515,Assiut, Assiut University
Other Study IDs: neonatal arrhythmias
Record Dates: First submitted 2024-09-11; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Neonatal Arrhythmias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
assess the Management and clinical outcome of neonatal arrhythmia

DETAILED DESCRIPTION:
Cardiac arrhythmia is a significant cardiovascular disorder in the neonatal period and can result in infant mortality if not diagnosed or treated promptly. The incidence of arrhythmia is about 0.1% to 4.8% during the neonatal period. In neonatal intensive care units (NICUs), the incidence of cardiac arrhythmia could reach 10%. Approximately 1% to 3% of fetal

* cardiac arrhythmias were detected during pregnancy The clinical presentation of NA is variable. Some neonates do not become symptomatic, and could not be diagnosed during
* neonatal period, whereas others may develop signs of congestive heart failure and cardiogenic shock even before birth The most common significant arrhythmia is supraventricular tachycardia (SVT), but atrial flutter (AFL), various forms of atrioventricular block (AVB), and ventricular tachycardia (VT) may also occur. Because of the immature physiology of
* the fetal and neonatal myocardium, heart failure may occur at either abnormally low or high ventricular rates

  * The electrocardiogram (ECG) is the gold standard for identifying problems with heart rate and regularity. However investigations of arrhythmias were hampered by their transitory nature. Monitoring rhythm patterns over extended duration makes Holter monitors a very helpful complementary noninvasive tool in the diagnosis of cardiac arrhythmias. It allows the cumulative evaluation of heart rhythm and rhythm variability, which is important in diagnosing silent and episodic
* arrhythmias in high-risk groups Medical management of SVT consists of a trial of vagal maneuvers, adenosine, and medications to maintain sinus rhythm such as beta blockers and class I or class III antiarrhythmic medications. For neonates who have hemodynamically

  * significant SVT, frequent SVT requiring medical management, pre-excitation on ECG, or congenital cardiac defect chronic medical treatment is appropriate. AF is common in newborns, usually in structurally normal hearts, and long term medical therapy besides initial conversion to sinus rhythm is usually not needed, given the low probability of recurrence
* the prognosis depends on the early recognition and proper management of the condition in some serious neonatal cases Precise diagnosis with risk stratification of patients with non-benign neonatal arrhythmia is needed to reduce morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Neonates up to 28 day with arrhythmia except premature atrial contraction.

Exclusion Criteria:

* More than 28 day
* Neonates with other diseases other than arrhythmia .

Ages: 1 Day to 28 Days | Sex: All
Age Groups: Child
Study Population: assess theIncidence, .Management and clinical outcome of neonatal arrhythmia .
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment | Baseline
  Assessment of clinical outcomes of neonatal arrhythmias at Assiut University Children's Hospital , If cases will die or become completely free or survive with some problems and if become on treatment or not
Management of arrhythmias | Baseline
  Management of neonatal arrhythmias in Assiut University Children's Hospital based on ECG and lab investigation

SECONDARY OUTCOMES:
Investigation | Baseline
  (12- lead ECG including three lead rhythm strip)
  * Insure that the rhythm and QTC will be calculated.
  * Checking urea and electrolytes, serum calcium, magnesium and blood sugar.
  * ECHO Cardioghraphy will be considered if there is a suspension on Clinical examination of structural Congenital Heart disease (mummer, absence of femoral pulse).
  * It will also be considered if there are frequent ventricular premature couplet.
  * Any infant who is symptomatic for Congenital or cyanotic cardiac disease or congestive cardiac failure will be immediately admitted to the neonatal unit and managed according to their clinical condition

REFERENCES:
- [Background] Na J, Wu S, Chen L, Qi Y, Yuan Y, Feng G, Wang X, Hei M. Clinical Outcomes and Medical Burdens of Neonatal Arrhythmias in Children's Hospitals in China: A Protocol for Multi-Center Retrospective Cohort Study. Pediatr Cardiol. 2024 Apr;45(4):814-820. doi: 10.1007/s00246-024-03421-z. Epub 2024 Feb 19. PMID 38374353
- [Background] Kundak AA, Dilli D, Karagol B, Karadag N, Zenciroglu A, Okumus N, Dogan V, Uzunalic N. Non benign neonatal arrhythmias observed in a tertiary neonatal intensive care unit. Indian J Pediatr. 2013 Jul;80(7):555-9. doi: 10.1007/s12098-012-0852-3. Epub 2012 Oct 4. PMID 23054850
- [Background] Badrawi N, Hegazy RA, Tokovic E, Lotfy W, Mahmoud F, Aly H. Arrhythmia in the neonatal intensive care unit. Pediatr Cardiol. 2009 Apr;30(3):325-30. doi: 10.1007/s00246-008-9355-4. Epub 2009 Jan 30. PMID 19184182